### NCT02228499

Title: Academic Achievement in Children with Asthma

Date: June 22, 2018

#### **Academic Achievement in Children with Asthma**

#### Abstract

Background: Asthma is the most common chronic disease of childhood with a prevalence that is 1.6 times greater in African American (AA) children than in Non-Hispanic White children. Nationally, 700,000 children are seen for asthma in Emergency Departments (ED) every year, which are seen at Children's National Health System (CN) in Washington, DC. School performance and school attendance has not been well studied in urban children with asthma, especially at the middle school level.

Objective: Our purpose is to test the hypothesis that children with asthma have worse school performance than middle school children without asthma in Washington DC public schools.

Methods: We will conduct a cross-sectional observational study of children in 3<sup>rd</sup>-8<sup>th</sup> grade in the 2015-2016 academic year with and without asthma recruited from the Emergency Departments and the IMPACT DC asthma clinic at CN. We will collect demographic information, asthma severity information (for cases), and request that parents mail report cards and standardized test scores directly to the investigators. We will use multivariable linear and logistic regression to determine if the presence of asthma is associated with school performance.

#### Research Plan

#### A. Background and Specific Aims

Asthma is the most common chronic disease of childhood with a prevalence that is 1.6 times greater in African American (AA) children than in Non-Hispanic White children.<sup>1</sup> Nationally, 700,000 children are seen for asthma in Emergency Departments (ED) every year, 1% of which are seen at Children's National Medical Center (CN) in Washington, DC. The asthma prevalence rate among African America (AA) children and teens in Washington, DC is 20% higher than the national rate<sup>2</sup> and overall ED utilization rates for asthma are 4.3 times the national rate.<sup>3</sup> In 2007, approximately 10.5 million school days were lost due to asthma.<sup>1</sup>

Asthma severity may impact academic performance due to increased absenteeism. A study of Canadian school children showed that children with the most severe asthma had the lowest math and reading scores.<sup>4</sup> Tsakiris also showed that children with asthma on inhaled corticosteroids had better academic achievement than children with asthma not on long-term controller therapy, suggesting that poor control is associated with worse school performance.<sup>5</sup>

However, academic performance is dependent on many other factors, such as socio-economic status of the local district and resources available. Availability of skilled nursing differs between schools, impacting children with asthma; Hillemeier's study of children with asthma in Pennsylvania schools showed that less than half of secondary schools had adequate school nurse coverage, and that this reduced services provided to children with asthma. Children whose asthma is not managed at school may be absent more often. Parental education also plays a part in a child's school performance. Tsakiris et al, showed that in Greece, lower parental education level was independently associated with poor school performance in children with asthma.

Early adolescence (ages 10-13) is identified as a time of great transition with both developmental and biologic changes; in this time period male children with asthma generally improve and female with asthma develop worsening asthma, likely due to hormone effects. It has been shown that programs to reduce asthma symptoms in both younger children (elementary school) and older children (high school) do not work well in early adolescent children (middle school).<sup>7</sup>

In addition, despite the National Asthma Education Prevention Program (NAEPP, 2007) guidelines that encourage the assessment of the quality of life (QOL) in children, there has been minimal research on QOL in children with asthma.

Given the scarcity of information on the association between pediatric asthma and academic achievement, school attendance, and the QOL, and the need to establish baselines within individual communities, we have designed a study to examine the association between asthma in children in grades 3-8 and academic achievement, school attendance, and the QOL. Our overall hypothesis is that children with asthma will have worse school performance compared to children without asthma.

**Specific Aim 1:** To determine the association between asthma and school performance by comparing grade point averages (GPA) in children from 3<sup>rd</sup>-8<sup>th</sup> grade with and without asthma. We will enroll an additional 60 children in grades 3-8 with asthma (cases) from the ED/IMPACT DC and compare them with a group of 60 children in grades 3-8 without asthma (controls) recruited from the ED. Report cards will be collected between May 2016-November 2016or until 60 cases and 60 controls have been recruited, and GPAs will be compared. We expect children with asthma will have lower GPAs .

В.

#### Significance:

School achievement in elementary and middle school students with asthma is not well understood; this study will be pivotal in identifying if middle school students with asthma in the Washington DC are performing more poorly than their non-asthmatic counterparts.

#### C. Preliminary studies

We have not previously studied academic success in children with asthma.

#### D. Research Design and Methods

We are proposing a cross-sectional case-control observational study of children in grades 3-8 to compare academic achievement and school attendance between children with and without asthma. 60 children with asthma (cases) will be recruited from the IMPACT DC clinic and/or ED and 60 children without asthma (controls) will be recruited from the ED. Recruitment will occur from May 2016 through November 2016.

Inclusion criteria for cases include asthma diagnosed by a clinician for greater than 1 year with a history of exacerbation requiring systemic corticosteroids within the past 2 years. Controls will have no history of asthma. All children, cases and controls, must (1) be in grade level 3-8 in the 2015-2016 school year, attend public school in Washington, DC (DCPS) and reside in their school district;(2) be accompanied by their parent or legal guardian. Exclusion criteria for cases and controls will be (1) presence of a chronic medical condition other than asthma or (2) a family that does not speak English or Spanish.

#### **Demographic Data for Cases and Controls**

Demographic information will be obtained by a structured interview; the questionnaire (Appendix A) will be used on both cases and controls: the parent/caregiver will be asked about the child's age, gender, race/ethnicity, insurance type. health care utilization, medications usage, highest level of education of the parent/ caregiver, income of the household, and parental report of school services. Cases will complete an additional 11 questions to determine asthma severity to determine NAEPP score and the Asthma Control Test (ACT) score (Appendix F and G).

We will utilize the child's electronic medical record (Cerner for ED charts and eClinicalWorks for the IMPACT DC charts) to determine insurance type and health care utilization. We will also determine each participant's weight and height from the medical record and will access medical records for the period of time we are collecting report cards for to determine clinical information, such as number of ED visits and hospitalizations over the 14 month period that the report cards cover (August 2015-November 2016).

#### Reporting of Academic Achievement and School Attendance

At the time of recruitment, families will be given a self-addressed, stamped envelope to send the child's 2013 first term (if available), standardized test score report (if available), and final report card to the research team. All report cards/score reports will be returned to the family via US Mail. Academic achievement, standardized test scores, and school attendance will be recorded from the report cards. All report cards in the DCPS system use the same grading scale..

#### **The Self-Perception Profile**

The self-perception profile is a reliable validated 6 question questionnaire for children in grades 6-8 that allows a child to self-evaluate their feelings about their engagement in school and their own school performance.

#### Reporting of the Quality of Life using the Peds QL 4.0 Form

QOL will be measured using the validated PedsQL 4.0 for children, teens, and parents (Appendices B, C, D, and E). The PedsQL 4.0 has four scales with 23 questions which ascertain physical functioning, emotional functioning, social functioning, and school functioning. A 5-point Likert scale is used in the child self-report and for the parent proxy reports. Items are reverse scored and linearly transformed to a 0 to 100 scale (0=100, 1=75, 2=50, 3=25, and 4=0), so higher scores indicate better QOL.

**E. Statistical analysis** Descriptive statistics will be used to analyze demographic variables (rates, proportions, means, medians, ranges). Univariate comparisons will be performed using appropriate categorical or continuous statistical analyses. Multivariate testing will be performed using logistic and/or liner regression where appropriate.

Sample Size: The study will be powered on the proportion of patients in each group with a grade point average >3.0. The overall proportion of DC public middle school students in the 2012-2013 school year with a GPA >3.0 was approximately 35%. Assuming that this figure is similar for children without asthma (controls), we will need 70 cases and 70 controls to have 80% power detect a 20% absolute difference in the proportion of children with asthma (cases) with a grade point average >3.0 (alpha = 0.05, two-sided).

We have chosen to include 120 children in the expansion of this original study, as we expect that less than 50% of all included patients will return their final year report cards via the self-addressed, stamped envelope.

#### F. Human Subjects

A convenience sample of potential participants' guardians will be approached in the temporal sequence that they are available either in the emergency department or in the IMPACT DC Asthma Clinic, informed about the research study, and invited to participate. Informed consent will obtained from all guardians.

After obtaining informed consent, trained research assistants and/or the investigators will use extant hospital electronic data and information obtained from questionnaires as the source of research material for this study.

- The risks of this study include inadvertent disclosure of protected health information. This risk does not exceed the daily risk of inadvertent disclosure of patients' protected health information during ED operations where patients' records are accessed through the ED tracking system of Logicare and the electronic medical records of EPRS.
- 2. There is the risk of feeling uncomfortable during the questionnaires; families will be told that some of the questions may make them uncomfortable and they are welcome to leave the study at any time, without penalty, if they feel uncomfortable. Alternatively, they may choose to leave questions unanswered.
- 3. There are no direct benefits to study participants. However, the knowledge gained from this study may allow us to identify a cohort of patients at special risk, for whom a targeted intervention would be appropriate.

4. Therefore, the risks are reasonable in relation to the benefits.

## G. Risks and Side Effects Questionnaires

Participants may find some of the questionnaires too personal; they will be offered the opportunity to refuse to answer any questions that make them feel uncomfortable. There is also the risk of breach of confidentiality; all participants will be assigned a random study number. This study number will be used to identify all questionnaires. Coding for the study numbers will be secured on a password protected file on the PI's hospital-issued laptop and stored on the secure CNMC server. We will store the study data in locked cabinets or offices.

#### H. Benefits

There are no direct benefits to participants.

#### I. Outside Consultants/Collaborators

None.

#### J. Contractual Agreements

None.

#### K. Costs To Subjects:

There is no cost to subjects.

#### L. Conflicts Of Interest:

There are no conflicts of interest.

#### M. Confidentiality:

The investigators will use reasonable measures to assure the security of these data, including locked office doors and file cabinets where paper records are stored, and secure, password-protected, computer software systems where electronic data are stored. The major risks to patients are the risks to confidentiality by inadvertent disclosure of protected health information. All paper data will be kept in the PI's locked office in locked file cabinets, to which only the PI will have keys for. All protected health information will be secured in password protected databases on the hospital Emergency Medical and Trauma Center (EMTC) drive. All research data will be de-identified and coded to further protect patient confidentiality. Code numbers and they respective medical record numbers will be kept in a separate password-protected database on the hospital's EMTC server. Passwords will only be known to the PI. These risks are reasonable in relation to the future anticipated benefits, which include identifying a future cohort of patients who might benefit from targeted interventions. The risk of inadvertent disclosure of protected health information is no more than minimal and no more than encountered on any patient visit to the ED.

#### N. Subject Compensation:

There will be no compensation for subjects on the expanded continuing portion of this study.

#### O. Facilities and Equipment

Existing departmental facilities will be used.

#### P. References & Literature Cited

- **1.** Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. *Pediatrics*. Mar 2009;123 Suppl 3:S131-145.
- 2. Moorman JE, Rudd RA, Johnson CA, et al. National surveillance for asthma--United States, 1980-2004. *MMWR Surveill Summ*. Oct 19 2007;56(8):1-54.
- **3.** Teach SJ. <u>www.impact-dc.org</u>. 2010.
- **4.** Kohen DE. Asthma and school functioning. *Health reports*. Dec 2010;21(4):35-45.
- **5.** Tsakiris A, Iordanidou M, Paraskakis E, et al. The presence of asthma, the use of inhaled steroids, and parental education level affect school performance in children. *BioMed research international*. 2013;2013:762805.
- **6.** Hillemeier MM, Gusic ME, Bai Y. Rural and urban children with asthma: are school health services meeting their needs? *Pediatrics*. Sep 2006;118(3):1097-1103.
- 7. Clark NM, Dodge JA, Thomas LJ, Andridge RR, Awad D, Paton JY. Asthma in 10- to 13-year-olds: challenges at a time of transition. *Clin Pediatr (Phila)*. Oct 2010;49(10):931-937.

Appendix A



| | Case# | |
|---|---|---|
| Understanding the Impact of Asthma in Academic Achieven | nent, School | Attendance, and |
| in the Quality of Life in Middle school aged child | ren Question | naire |

#### **Baseline Measure**

These questions will ask about your child's background and asthma history. In order for this study to be useful for families of children with asthma, it is important that everyone give us accurate answers. IMPACT DC team members will not share or discuss any personal information without your permission.

If you have any questions, please let me know. If not, we can start.

#### \*\*Note to Interviewers:

- Bold scripting is meant to be read to participants.
- [Italicized in brackets] scripting is a note for clarification that is not meant to be read aloud.

| General Information | |
|---|---|
| Interviewer's Initials | |
| Interview Date | /(mm/dd/yy) |
| Time of Interview Start | : [based on 24-hr clock] |
| Patient's Initials | |
| Patient's Date of Birth | /(mm/dd/yyyy) |
| Patient's Gender | Male Female |
| Which grade did your child complete in the | last 12 months at school |
| Two best contact phone numbers | and |
| Best contact Address | |
| Health Care Utilization | |
| - | hospitals other than Children's National on ional Emergency Room at the United Medical |
| In the last 12 months, have you been to an<br>Emergency Room at either Children's Natio | Emergency Room other than the Children's nal or the United Medical Center? |
| 1. No [Skip to next section] | |
| Yes [go to question 5] | |
| | 2 months has (CHILD) been to an Emergency<br>n's Emergency Room at either Children's National or |
| | 2 months has (CHILD) been admitted to a hospital al Medical Center for asthma? |

| 4. | How many times in the last 12 months has (CHILD) been in the PICU (Pediatric Intensive Care Unit) of a hospital other than Children's National Medical Center? |
|---|---|
| | times |
| Current Medic | cation Use |
| actual respons<br>medicines. If i | ptions for types of medicines. Just read question as worded, and then record se and classify medication. <u>Do not</u> show pictures or demos/samples of asthma name unknown but respondent describes medication, or medication is unknown, ual response and classify as "Other".] |
| 5. | During the past two days, did [CHILD] take or use any medications including pills, syrups, or inhaled medications? |
| | Yes No [skip to question 6) Don't know [skip to question 7) |
| If y | es: |
| | Which medicines? |
| | Andhor a Nandinaking a |
| | Asthma Medications: |
| | Inhaled or nebulized steroid (ex. Pulmicort, Flovent, QVAR, Asmanex) |
| | Short-acting bronchodilator (ex. albuterol, Ventolin, ProAir, Xopenex) |
| | Long-acting bronchodilator (ex. salmeterol, formoterol) |
| | Inhaled steroid/LABA combination (ex. Advair, Symbicort, Dulera) |
| | Long-acting leukotriene inhibitor (ex. Singulair) |
| | Oral Steroid (Prednisone, Prednisolone, Dexamethasone) |
| | Other: |
| | Allergy Medications: |
| | Antihistamines |
| | Intranasal Steroid |
| | Other: |
| | Non-asthma/allergy medication: |

#### Adherence:

| 6.<br>Ye | Does your child take a daily medicine? No [Skip to question 7] |
|---|---|
| | What is the name of this medication: |
| | Asthma Medications: |
| | Inhaled or nebulized steroid (ex. Pulmicort, Flovent, QVAR, Asmanex) |
| | Short-acting bronchodilator (ex. albuterol, Ventolin, ProAir, Xopenex) |
| | Long-acting bronchodilator (ex. salmeterol, formoterol) |
| | Inhaled steroid/LABA combination (ex. Advair, Symbicort, Dulera) |
| | Long-acting leukotriene inhibitor (ex. Singulair) |
| | Oral Steroid (Prednisone, Prednisolone, Dexamethasone) |
| | Other: |
| | Allergy Medications: |
| | Antihistamines |
| Other: | |
| Non-asthma/a | llergy medication: |
| Demographic | / Family History |
| Finally, resea | rch studies always ask a few questions about your family background. |
| 7. | What do you consider [CHILD]'s race to be? [Read options and circle all that apply] |
| Bla | ck or African-American |
| Asia | American Indian or Alaska Native |
| □Nat | ive Hawaiian/Pacific Islander Some other race: |
| | What do you consider [CHILD]'s ethnicity to be? [Read options] |

| ☐ Non-Hispanic |
|---|
| Other: |
| 8. Do any of [CHILD]'s parents, brothers, or sisters have asthma? [Include those who do and do not live in household.] |
| Yes Don't know |
| 9. How many days of school did you child miss over the last school year due to asthma? |
| 10. Does your child receive any special services at school? What are they? |
| 11. What is the highest grade or school level that you have completed? Never attended school |
| Grade 1-11 |
| ☐ GED or 12 <sup>th</sup> grade |
| Some college/technical/vocational training |
| College graduate |
| Other: |
| 12. Keeping in mind the various possible sources of income for your household, su |

12. Keeping in mind the various possible sources of income for your household, such as a job, supplemental security income (SSI) or disability, social security, public assistance, food stamps, unemployment compensation, and child support, what was the total income during [LAST CALENDAR YEAR] from all sources for everyone in your household? Please point to the answer closest to your total household income.

[Show categories listed on hand card. Ask for last full calendar year. If the respondent cannot give a figure, go over each source of income and get an estimate per month and multiply by twelve]

| \$5,000 or less | \$5,001 - \$10,000 | \$10,001 - \$20,000 |
|---|---|---|
| S20,001 - \$30,000 | \$30,001 - \$40,000 | \$40,001 - \$50,000 |
| S50,001 - \$60,000 | \$60,001 - \$70,000 | \$70,001 - \$80,000 |
| S80,001 - \$90,000 | \$90,001 - \$100,000 | \$100,001 - \$150,000 |
| S150,001 - \$200,000 | \$200,001 - \$250,000 | \$250,001 or greater |
| Refused | Don't know | |
| Thank you very much for answeri improve care for children with ast compensated with a \$25 gift card | hma. As we discussed earl | ier, you will be |
| [Caregiver given copy of info | rmed consent document] | |
| Time of Interview End | : [based on 2 | 24-hr clock] |
| Interviewer Comments | | |
| Please indicate if respondent had disprovided inaccurate or misleading resort the interview, or the respondent has specific questions if appropriate. | esponses, there were any unu | sual circumstances at the time |
| Chart Review | | |

[To be completed <u>after</u> visit in IMPACT DC Asthma Clinic is completed]

From IMPACT DC Clinic Form:

| 13. Final Asthma Classification [based on clinician's assessment] |
|---|
| ☐ Mild Persistent |
| Moderate Persistent |
| Severe Persistent |
| 14. Insurance type |
| 12a. Name of child's insurance provider: |
| 12b. Insurance type: |
| Public |
| Private |
| None |
| Unknown |
| 15. Zip code of residence: |
| 16. Oral Steroids: How many courses of oral steroids in the prior 12 months: |
| 17. If applicable: If a patient is already using an ICS, what was the number of puffs displayed on the back of the inhaler they are currently using? of puffs |
| From Medical Records: |
| Health Care Utilization [from medical records, visits to Children's Hospital or any of the Goldberg Center Children's Health Centers]: |
| Emergency Department visits for asthma |
| 18. Number of ED visits in prior 12 months: 19. Hospitalizations for asthma 20. Number of hospitalizations in prior 12 months: 21. PICU Admissions |

| Number of PICU admissions in the last 12 months: |
|---------------------------------------------------------------|
| 21.Urgent care visits for asthma (if Goldberg Center patient) |
| Number of urgent care visits in prior 12 months: |
| Appendix B |

# PedsQL Pediatric Quality of Life Inventory

Version 4.0

PARENT REPORT for CHILDREN (ages 8-12)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for **your child**.

Please tell us **how much of a problem** each one has been for **your child** during the **past ONE month** by circling:

**0** if it is **never** a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

### In the past ONE month, how much of a problem has your child had with

| PHYSICAL FUNCTIONING (problems with) | Never | Almos<br>t<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Walking more than one block | 0 | 1 | 2 | 3 | 4 |
| 2. Running | 0 | 1 | 2 | 3 | 4 |
| Participating in sports activity or exercise | 0 | 1 | 2 | 3 | 4 |
| 4. Lifting something heavy | 0 | 1 | 2 | 3 | 4 |
| 5. Taking a bath or shower by him or herself | 0 | 1 | 2 | 3 | 4 |
| 6. Doing chores around the house | 0 | 1 | 2 | 3 | 4 |
| 7. Having hurts or aches | 0 | 1 | 2 | 3 | 4 |
| 8. Low energy level | 0 | 1 | 2 | 3 | 4 |

| EMOTIONAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. Feeling sad or blue | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling angry | 0 | 1 | 2 | 3 | 4 |
| 4. Trouble sleeping | 0 | 1 | 2 | 3 | 4 |
| 5. Worrying about what will happen to him or her | 0 | 1 | 2 | 3 | 4 |
| SOCIAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
| Getting along with other children | 0 | 1 | 2 | 3 | 4 |
| 2. Other kids not wanting to be his or her friend | 0 | 1 | 2 | 3 | 4 |
| Getting teased by other children | 0 | 1 | 2 | 3 | 4 |
| 4. Not able to do things that other children his or her | 0 | 1 | 2 | 3 | 4 |
| 5. Keeping up when playing with other children | 0 | 1 | 2 | 3 | 4 |
| SCHOOL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
| Paying attention in class | 0 | 1 | 2 | 3 | 4 |
| 2. Forgetting things | 0 | 1 | 2 | 3 | 4 |
| Keeping up with schoolwork | 0 | 1 | 2 | 3 | 4 |

| Missing school because of not feeling well | 0 | 1 | 2 | 3 | 4 |
|---------------------------------------------------|---|---|---|---|---|
| 5. Missing school to go to the doctor or hospital | 0 | 1 | 2 | 3 | 4 |

Appendix C

# PedsQL Pediatric Quality of Life Inventory

Version 4.0 CHILD REPORT (ages 8-12)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for you.

Please tell us **how much of a problem** each one has been for you during the **past ONE month** by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers. If you do not understand a question, please ask for help.

In the past ONE month, how much of a problem has this been for you ...

| ABOUT MY HEALTH AND ACTIVITIES (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almos<br>Alway |
|---|---|---|---|---|---|
| It is hard for me to walk more than one block | 0 | 1 | 2 | 3 | 4 |
| 2. It is hard for me to run | 0 | 1 | 2 | 3 | 4 |
| 3. It is hard for me to do sports activity or exercise | 0 | 1 | 2 | 3 | 4 |
| 4. It is hard for me to lift something heavy | 0 | 1 | 2 | 3 | 4 |
| 5. It is hard for me to take a bath or shower by myself | 0 | 1 | 2 | 3 | 4 |
| 6. It is hard for me to do chores around the house | 0 | 1 | 2 | 3 | 4 |
| 7. I hurt or ache | 0 | 1 | 2 | 3 | 4 |
| 8. I have low energy | 0 | 1 | 2 | 3 | 4 |

| ABOUT MY FEELINGS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almos<br>Alway |
|---|---|---|---|---|---|
| I feel afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. I feel sad or blue | 0 | 1 | 2 | 3 | 4 |
| 3. I feel angry | 0 | 1 | 2 | 3 | 4 |
| 4. I have trouble sleeping | 0 | 1 | 2 | 3 | 4 |
| 5. I worry about what will happen to me | 0 | 1 | 2 | 3 | 4 |

| How I GET ALONG WITH OTHERS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almo<br>Alwa |
|---|---|---|---|---|---|
| I have trouble getting along with other kids | 0 | 1 | 2 | 3 | 4 |
| 2. Other kids do not want to be my friend | 0 | 1 | 2 | 3 | 4 |
| 3. Other kids tease me | 0 | 1 | 2 | 3 | 4 |
| 4. I cannot do things that other kids my age can do | 0 | 1 | 2 | 3 | 4 |
| 5. It is hard to keep up when I play with other kids | 0 | 1 | 2 | 3 | 4 |
| ABOUT SCHOOL (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almo:<br>Alway |
| It is hard to pay attention in class | 0 | 1 | 2 | 3 | 4 |
| | 1 | | | ! | 1 |
| 2. I forget things | 0 | 1 | 2 | 3 | 4 |
| <ul><li>2. I forget things</li><li>3. I have trouble keeping up with my schoolwork</li></ul> | 0 | 1 | 2 | 3 | 4 |
| | | 1 1 1 | | | |



# Version 4.0 PARENT REPORT for TEENS (ages 13-18)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for **your teen**.

Please tell us **how much of a problem** each one has been for **your teen** during the **past ONE month** by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

In the past ONE month, how much of a problem has your teen had with ...

| PHYSICAL FUNCTIONING (PROBLEMS WITH) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Walking more than one block | 0 | 1 | 2 | 3 | 4 |
| 2. Running | 0 | 1 | 2 | 3 | 4 |
| Participating in sports activity or exercise | 0 | 1 | 2 | 3 | 4 |
| 4. Lifting something heavy | 0 | 1 | 2 | 3 | 4 |
| 5. Taking a bath or shower by him or herself | 0 | 1 | 2 | 3 | 4 |
| 6. Doing chores around the house | 0 | 1 | 2 | 3 | 4 |
| 7. Having hurts or aches | 0 | 1 | 2 | 3 | 4 |
| 8. Low energy level | 0 | 1 | 2 | 3 | 4 |

| EMOTIONAL FUNCTIONING (PROBLEMS WITH) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. Feeling sad or blue | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling angry | 0 | 1 | 2 | 3 | 4 |
| 4. Trouble sleeping | 0 | 1 | 2 | 3 | 4 |
| 5. Worrying about what will happen to him or her | 0 | 1 | 2 | 3 | 4 |
| SOCIAL FUNCTIONING (PROBLEMS WITH) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
| Getting along with other teens | 0 | 1 | 2 | 3 | 4 |
| 2. Other teens not wanting to be his or her friend | 0 | 1 | 2 | 3 | 4 |
| Getting teased by other teens | 0 | 1 | 2 | 3 | 4 |
| 4. Not able to do things that other teens his or her age can do | 0 | 1 | 2 | 3 | 4 |
| 5. Keeping up with other teens | 0 | 1 | 2 | 3 | 4 |
| SCHOOL FUNCTIONING (PROBLEMS WITH) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
| Paying attention in class | 0 | 1 | 2 | 3 | 4 |
| 2. Forgetting things | 0 | 1 | 2 | 3 | 4 |
| Keeping up with schoolwork | 0 | 1 | 2 | 3 | 4 |
| 4. Missing school because of not feeling well | 0 | 1 | 2 | 3 | 4 |
| 5. Missing school to go to the doctor or hospital | 0 | 1 | 2 | 3 | 4 |

Appendix E

# PedsQL Pediatric Quality of Life Inventory

Version 4.0 **TEEN REPORT** (ages **13-18**)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for you.

Please tell us **how much of a problem** each one has been for you during the **past ONE month** by circling:

**0** if it is **never** a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

| ABOUT MY HEALTH AND ACTIVITIES (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| It is hard for me to walk more than one block | 0 | 1 | 2 | 3 | 4 |
| 2. It is hard for me to run | 0 | 1 | 2 | 3 | 4 |
| 3. It is hard for me to do sports activity or exercise | 0 | 1 | 2 | 3 | 4 |
| 4. It is hard for me to lift something heavy | 0 | 1 | 2 | 3 | 4 |
| 5. It is hard for me to take a bath or shower by myself | 0 | 1 | 2 | 3 | 4 |
| 6. It is hard for me to do chores around the house | 0 | 1 | 2 | 3 | 4 |
| 7. I hurt or ache | 0 | 1 | 2 | 3 | 4 |
| 8. I have low energy | 0 | 1 | 2 | 3 | 4 |

| ABOUT MY FEELINGS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| I feel afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. I feel sad or blue | 0 | 1 | 2 | 3 | 4 |
| 3. I feel angry | 0 | 1 | 2 | 3 | 4 |
| 4. I have trouble sleeping | 0 | 1 | 2 | 3 | 4 |
| 5. I worry about what will happen to me | 0 | 1 | 2 | 3 | 4 |
| How I GET ALONG WITH OTHERS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
| I have trouble getting along with other teens | 0 | 1 | 2 | 3 | 4 |
| Other teens do not want to be my friend | 0 | 1 | 2 | 3 | 4 |
| 3. Other teens tease me | 0 | 1 | 2 | 3 | 4 |
| 4. I cannot do things that other teens my age can do | 0 | 1 | 2 | 3 | 4 |
| 5. It is hard to keep up with my peers | 0 | 1 | 2 | 3 | 4 |
| ABOUT SCHOOL (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
| It is hard to pay attention in class | 0 | 1 | 2 | 3 | 4 |
| 2. I forget things | 0 | 1 | 2 | 3 | 4 |
| I have trouble keeping up with my schoolwork | 0 | 1 | 2 | 3 | 4 |
| 4. I miss school because of not feeling well | 0 | 1 | 2 | 3 | 4 |
| 5. I miss school to go to the doctor or hospital | 0 | 1 | 2 | 3 | 4 |

Appendix F



| Case# |
|-------|

Understanding the Impact of Asthma in Academic Achievement, School Attendance, and in the Quality of Life in Middle school aged children Questionnaire Using The NAEPP, 2007 guidelines

The next series of questions will ask about your child's severity of asthma, it is important that everyone give us accurate answers. The team members will not share or discuss any personal information without your permission. Only the other team members will be able to see your answers to questions or your name. Everything is kept private and strictly confidential. None of your answers will in any way affect your medical care, benefits, any services you may be receiving (such as Medicaid or WIC) or your job or immigration status. You can decide at any point not to participate in the study, and your decision won't have any impact on your current or future medical care. If you have any questions, please let me know. If not, we can start.

The next series of questions will ask about child's asthma over the past 2-4 weeks. Please listen to all the possible responses and then pick the one that best describes the child situation. You must pick the single best answer that describes the childs situation over the prior 2-4 weeks.

So think about the last 2-4 weeks....

| 1how often during the day did | have asthma symptoms? |
|-------------------------------|-----------------------|
|-------------------------------|-----------------------|

| 5-11 years | | | |
|---|---|---|---|
| | Severity | | Control |
| а | <2d/wk | а | < 2d/wk but not > 1x/d |
| b | >2d/wk but not daily | b | >2d/wk or many<br>times on< 2d/wk |
| С | Daily | | |
| d | Throughout the day | С | Throughout the day |

| | ≥ 12 years | | |
|---|----------------------|---|-----------------------------------|
| | Severity | | Control |
| а | <2d/wk | а | < 2d/wk but not > 1x/d |
| b | >2d/wk but not daily | b | >2d/wk or many<br>times on< 2d/wk |
| С | Daily | | |
| d | Throughout the day | С | Throughout the day |

| 2 | .how often during | the night did | awake due to asthma symptoms? |
|---|---|---|---|
| <b>4</b> | .IIOW OILEII GUIIIIG | LIIG IIIUIIL UIU | awake due to astillia syllibtollis: |

| 5-11 years | | | |
|------------|------------------------|---|------------|
| | Severity | | Control |
| а | <2x/month | а | 0-1x/month |
| b | 3-4 x/month | b | >2x/month |
| С | >1x/wk but not nightly | С | ≥2x/wk |
| d | Often 7x/wk | | |

| ≥ 12 years | | | |
|------------|------------------------|---|-------------------|
| | Severity | | Control |
| а | <2x/month | а | < 2x/month |
| b | 3-4 x/month | b | 1-3x/wk |
| С | >1x/wk but not nightly | С | <u>&gt;</u> 4x/wk |
| d | Often 7x/wk | | |

3...how often during the night did \_\_\_\_\_use albuterol, quick relief medicines, for asthma symptoms? (please do not include albuterol before exercise or heavy play to avoid wheezing due to exercise).

| | 5-11 years | | |
|------------------|----------------|---|-------------|
| Severity Control | | | |
| а | <2d/wk | а | < 2d/wk |
| b | >2d/wk but not | b | >2d/wk |
| | daily | | |
| С | Daily | | |
| d | several x/d | С | several x/d |

| | ≥ 12 years | | |
|---|----------------|---|----------------|
| | Severity | | Control |
| а | <2d/wk | а | < 2d/wk |
| b | >2d/wk but not | b | >2d/wk |
| | daily | | |
| С | Daily | | |
| d | Several x/d | С | Throughout the |
| | | | day |

#### 4...how often did asthma interfere with the childs normal activity.

| 5-11 years | | | |
|------------------|------------------|---|-----------------|
| Severity Control | | | |
| a | None | a | none |
| b | minor limitation | b | some limitation |

| С | some limitation | | |
|---|-------------------|---|-------------------|
| d | extremely limited | С | extremely limited |

| <u>&gt;</u> 12 years | | | |
|----------------------|-------------------|---|-------------------|
| Severity Control | | | |
| а | None | а | none |
| b | minor limitation | b | some limitation |
| С | some limitation | | |
| d | extremely limited | С | extremely limited |

5...Now I need to know how many separate times child took steroids by mouth over the last year to treat an asthma attack. A steroid by mouth is a pill or syrup that is taken for a short period of time to treat asthma attacks.

| 5-11 years | | | |
|------------------|---------------|---|---------------|
| Severity Control | | | |
| а | 0-1/last year | а | 0-1/last year |
| b | >2x last year | b | 2xlast year |

| ≥12 years | | | |
|-----------|---------------|---|---------------|
| | Severity | | Control |
| а | 0-1/last year | а | 0-1/last year |
| b | ≥2x last year | b | 2xlast year |

### Appendix G



| IMP | <b>ACT</b> | <b>C</b> | | | |
|---|---|---|---|---|---|
| Improving Pediatric Asth | ma Care in the District of Columbia | ~ | Case# | | |
| <b>in the Quali</b> t<br>The American L<br>ControlTest, no | ty of Life in Mide<br>ung Association reco<br>matter how well co<br>core that may help y | <b>dle school aged c</b><br>ommends everyone 12<br>ontrolled you think you | hildren<br>2 years of age and older<br>1r asthma is. Your answ | nt, School Attendance<br>r with asthma take the Asth<br>yers to this 5-question quiz<br>tent plan is working or if it | nma<br>will |
| How to take the | e Asthma Control Te | st | | | |
| Step 1. Write th | ne number of each a | nswer in the score box | provided. | | |
| Step 2. Add up | each score box for y | our total. | | | |
| Step 3. Take the | e test to your doctor | to talk about your tot | al score. | | |
| 1.In the past 4 or at home? | weeks, how much of | the time did your astl | nma keep you from get | ting as much done at work | , scho |
| all the time<br>1 | most of the time<br>2 | some of the time | a little of the time<br>4 | None of the time<br>5 | |
| 2.During the pa | st 4 weeks, how ofto | en have you had short | ness of breath? | | |
| More than once a day | Once a day | 3-5 times a week | Once or twice a<br>week<br>4 | Not at all | |
| 3.During the pa | | | mptoms (wheezing, cou | ghing, shortness of breath | L<br>, ches |
| 4 or more<br>nights a week | 2-3 nights a week | once a week | once or twice | Not at all | |
| 1 | 2 | 3 | 4 | 5 | |
| 4.During the paalbuterol)? | st 4 weeks,how ofte | n have you used your | rescue inhaler or nebu | ılizer medication (such as | |
| 3 or more time<br>per day<br>1 | s 1-2 times<br>per day | 2-3 times per week<br>3 | once a week or less<br>4 | Not at all | |
| | | control during thepas | t 4 weeks? | ı | |
| | | T | 1 | | |

| not controlled at all | poorly<br>controlled | somewhat controlled | well controlled | completely controlled |
|---|---|---|---|---|
| 1 | 2 | 3 | 4 | 5 |

Appendix H
Conversation Guide with Participants

Thank you for completing the questionnaires, would you please provide your two best phone numbers so that we may contact you and your best contact mailing address. I have also provided you with an addressed and stamped envelope for you to mail your child's report card to me. We will send you a \$25.00 gift card from Target when we receive your child's report card and we will return you child's report card once we have abstracted the information we need.

#### References:

- **1.** Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. *Pediatrics*. Mar 2009;123 Suppl 3:S131-145.
- 2. Moorman JE, Rudd RA, Johnson CA, et al. National surveillance for asthma--United States, 1980-2004. *MMWR Surveill Summ.* Oct 19 2007;56(8):1-54.
- **3.** Teach SJ. www.impact-dc.org. 2010.
- **4.** Kohen DE. Asthma and school functioning. *Health reports*. Dec 2010;21(4):35-45.
- **5.** Tsakiris A, Iordanidou M, Paraskakis E, et al. The presence of asthma, the use of inhaled steroids, and parental education level affect school performance in children. *BioMed research international*. 2013;2013:762805.
- **6.** Hillemeier MM, Gusic ME, Bai Y. Rural and urban children with asthma: are school health services meeting their needs? *Pediatrics*. Sep 2006;118(3):1097-1103.
- 7. Clark NM, Dodge JA, Thomas LJ, Andridge RR, Awad D, Paton JY. Asthma in 10- to 13-year-olds: challenges at a time of transition. *Clin Pediatr (Phila)*. Oct 2010;49(10):931-937.